CLINICAL TRIAL: NCT01698034
Title: How Volunteer Programs Affect Health and Well-being in Low-income Youth
Brief Title: Volunteering and Cardiovascular Risk in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: William T. Grant Foundation (Other); HopeLab Foundation (Other); Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H11-00943
Record Dates: First submitted 2012-09-21; First posted 2012-10-02 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Cardiovascular Risk Factors
Keywords: volunteering; cardiovascular health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Volunteering (Experimental): Weekly volunteering with elementary school children in after school programs
  Interventions: Behavioral: Volunteering
- Control (No Intervention): Wait-list control

INTERVENTIONS:
Behavioral: Volunteering — Weekly volunteering with elementary school children in after school programs
  Arms: Volunteering

SUMMARY:
This study tested whether getting youth engaged in helping others (volunteering) would benefit youth's physical health. 106 predominantly minority and low socioeconomic status (SES) youth were randomized to either volunteer weekly with elementary school children in after school programs or to a wait-list control group. The investigators hypothesized that cardiovascular risk markers of C-reactive protein (CRP), interleukin-6 (IL-6), total cholesterol, and body mass index (BMI) would be lower at post-intervention (4 months after baseline) in the volunteer group compared to the control group. The investigators also hypothesized that the intervention might work through pathways such as reducing negative mood, improving self esteem, and increasing prosocial behaviors (empathy, altruism).

ELIGIBILITY:
Inclusion Criteria:

* 10th grade high school student
* English speaking
* No chronic illnesses

Exclusion Criteria:

* Chronic medical illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Body mass index | Baseline-adjusted post-intervention scores at 4 months
C-reactive protein | Baseline-adjusted post-intervention scores at 4 months
Interleukin-6 | Baseline-adjusted post-intervention scores at 4 months
Total Cholesterol | Baseline-adjusted post-intervention scores at 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Edith Chen, Principal Investigator — Northwestern University
Locations (1):
- Vancouver Technical Secondary School, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Schreier HM, Schonert-Reichl KA, Chen E. Effect of volunteering on risk factors for cardiovascular disease in adolescents: a randomized controlled trial. JAMA Pediatr. 2013 Apr;167(4):327-32. doi: 10.1001/jamapediatrics.2013.1100. PMID 23440253